CLINICAL TRIAL: NCT04776681
Title: Living With Marfan Syndrome II: the Psychosocial and Health-related Quality of Life Effects of Surgical Interventions for Aorto-vascular Manifestations (LIMA II Study)
Brief Title: Living With Marfans and Your Aorta: Surgical Outcomes Study
Acronym: LIMA II
Status: Recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Aortic Dissection Awareness UK & Ireland. (Other)
Responsible Party: Sponsor
Other Study IDs: 293099
Record Dates: First submitted 2021-02-18; First posted 2021-03-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Marfan Syndrome; Marfan Syndrome Cardiovascular Manifestations
MeSH Terms: conditions — Marfan Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Marfan Syndrome (MFS) is a genetic disease affecting the eyes, skeleton, heart and arteries. Despite MFS affecting multiple organ systems, cardiovascular manifestations are the most serious and life threatening. Approximately 80% of adult MFS patients will have a dilated aortic root by age 40 years with aortic aneurysm and dissection the leading causes of morbidity and mortality. Living with a diagnosis of Marfan Syndrome, including undergoing and recovering from heart surgery, affects patients' mental health, well-being and quality of life in ways that are not well understood.

This study will address the current knowledge gaps in this area and will provide the information needed to design interventions to help improve the MFS patients' mental health, well-being and quality of life after heart surgery. The study will include adult MFS patients who are undergoing aorto-vascular surgery.

The overall aim of the study is to explore the psychosocial and health-related quality of life (HRQoL) effects of the surgical interventions for aorto-vascular manifestations of MFS in 3 large UK cardiac centres. To achieve this, the researchers will ask the potential participants, after obtaining informed consent, to complete a series of accepted / validated questionnaires to measure the health-related quality of life (SF-36 and EQ5D questionnaire) and psychosocial factors such as depression (CES-D questionnaire), fatigue (Fatigue Severity Scale), stigma (Perceived Stigma Questionnaire), self-esteem (Rosenberg Self-esteem Scale), pain and illness perception (Illness Perception Questionnaire). Participants will be asked to complete the questionnaires before surgery and at various time points after surgery (at 6 weeks after hospital discharge and at 6 and 12 months after surgery). The research team will also collect in-hospital post-operative morbidity burden following aorto-vascular surgery using cardiac post-operative morbidity score (C-POMS) tool from the patients and clinical records. The association of C-POMS with psychosocial and HRQoL outcomes will also be examined.

DETAILED DESCRIPTION:
Marfan Syndrome (MFS) is a rare autosomal-dominant connective tissue disorder with pleiotropic manifestations primarily affecting the skeletal, ocular, and cardiovascular systems. Despite MFS affecting multiple organ systems, cardiovascular manifestations are the most serious and life threatening. Approximately 80% of adult MFS patients will have a dilated aortic root by age 40 years with aortic aneurysm and dissection the leading causes of morbidity and mortality. However, there is limited evidence worldwide on health-related quality of life (HRQoL) and psychosocial aspects of the recovery of MFS patients undergoing surgical intervention. Undergoing a heart operation can be a stressful and life-threatening experience involving a lot of uncertainties, long periods of absence from work and social activities as well as limitation on physical activities which can potentially lead to psychosocial problems and poor health-related quality of life. Therefore, there is a specific need for high quality descriptive and exploratory research in this area.

The overarching aim of this prospective observational cohort study is to explore the psychosocial and HRQoL effects of surgical interventions for aorto-vascular manifestations of MFS in three large UK cardiac centres. Potential participants will be recruited from the outpatient pre-admission clinic. HRQoL and psychosocial factors will be determined and quantified using validated questionnaires before surgery and at various time points after surgery (at 6 weeks after hospital discharge and at 6 and 12 months after surgery). The questionnaires will be delivered either in paper or electronic format, depending on participant's preference. In-hospital post-operative morbidity burden following aorto-vascular surgery using cardiac post-operative morbidity score (C-POMS) tool will also be determined from the patients and clinical records and its association with psychosocial and HRQoL outcomes will be examined.

The outcome of the study will significantly contribute to the UK and international evidence-base on the HRQoL and psychosocial impact of the aorto-vascular surgical interventions on MFS patients and will provide clinicians with the foundation that will serve as basis for appropriate interventions. The result will also be useful to better understand the condition and potentially guide the researchers in devising a patient care pathway that includes this aspect of care as well as develop a holistic and comprehensive service for this patient group.

ELIGIBILITY:
Inclusion Criteria:

1. >/= 18 years old at the time of surgery;
2. have validated diagnosis of MFS (using revised Ghent criteria);
3. having aorto-vascular surgery

Exclusion Criteria:

1. <18years old at the time of surgery
2. Unable or unwilling to give written informed consent.
3. Inability to understand written and/or verbal English

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible consecutive patients with a diagnosis of MFS at three large UK cardiac centres will be identified prior to surgery, either through pre-operative outpatient clinic or via the clinical team.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Health-related Quality of Life (HRQoL) | before surgery, 6 weeks after hospital discharge, 6 months and 12 months after surgery
  HRQoL will be measured using the Short Form Health Survey 36 (SF-36). SF-36 consists of 8 sub-scales. All scales do contribute in different proportions to the scoring of the physical and mental dimensions, represented by the Physical Component Summary (PCS) and Mental Component Summary (MCS). Using an algorithm, raw scores can be converted to a transformed scale scores ranging from 0-100, with higher score indicating a better health state.
Change from Baseline Health-related Quality of Life (HRQoL) | before surgery, 6 weeks after hospital discharge, 6 months and 12 months after surgery
  HRQoL will be measured using EQ-5D. EQ-5D is divided into 2 components: health care description and evaluation. In the description part, summation of score ranges from 1 to 3; with 1 indicates the best health state and 3 indicates more severe or frequent problem. The evaluation part utilises a visual analogue scale to indicate the general health status with 100 indicating the best health status and 0 indicating the worst health status.

SECONDARY OUTCOMES:
Change from baseline psychosocial factor: depression | before surgery, 6 weeks after hospital discharge, 6 months and 12 months after surgery
  Depression will be measured using Centre for Epidemiological Studies Depression Scale (CES-D). The overall score ranges from 0 to 60, with higher scores indicating a more severe depressive symptoms. In general population, a cut-off score of 16 or above is used to identify those with significant clinical signs of depression.
Change from baseline psychosocial factor: fatigue | before surgery, 6 weeks after hospital discharge, 6 months and 12 months after surgery
  Fatigue will be determined using Fatigue Severity Scale (FSS). The minimum possible score is 9 and maximum possible score is 63. Higher score indicates greater fatigue severity.
Change from baseline psychosocial factor: stigma | before surgery, 6 weeks after hospital discharge, 6 months and 12 months after surgery
  Stigma will be measured using Perceived Stigma Questionnaire (PSQ). PSQ is composed of 4 sub-scales. Score on each sub-scale ranges from 1 to 6. Mean scores of >/= 2.0 on the devaluation and discrimination sub-scale indicates feeling of discriminated against or devalued. Mean scores of </= 3.5 on the withdrawal and secrecy sub-scales and </= 2.0 on the education sub-scale indicates the use of secrecy / withdrawal and education as coping styles, respectively.
Change from baseline psychosocial factor: self esteem | before surgery, 6 weeks after hospital discharge, 6 months and 12 months after surgery
  Self-esteem will be measured using Rosenberg Self-esteem Scale (RSS); score ranges from 10 (min) -40 (max); higher score indicates higher self-esteem.
Change from baseline psychosocial factors: pain and illness perception | before surgery, 6 weeks after hospital discharge, 6 months and 12 months after surgery
  Pain and Illness Perception will be determined using Illness Perception Questionnaire (IPQ). IPQ is divided into 5 components. The identity component is scored by summing the number of items identified at 'occasionally' or greater resulting to a total score ranging from 0 to 12 for the core list. The four other components are presented in mixed order and can be rated using a 5-point Likert scale ranging from 'strongly disagree' (1) to 'strongly agree (5).
Change from baseline post-operative morbidity outcomes | 3, 5, 8 and 15 days after surgery
  In-hospital post-operative morbidity outcomes will be identified and quantified using the Cardiac Post-Operative Morbidity Score (C-POMS) tool. C-POMS is a simple, validated tool assessing in-hospital total morbidity burden (score 0-13) derived by noting the presence of 13 morbidity domains on days three (D3), five (D5), eight (D8) and fifteen (D15) after surgery. Higher scores indicate more in-hospital post-operative morbidity.

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomews Hospital, London, United Kingdom